CLINICAL TRIAL: NCT05405439
Title: Phase Ib/II Clinical Study of TQB3823 Tablets Combined With Abiraterone Acetate Tablets and Prednisone Acetate Tablets in Patients With Metastatic Castration-resistant Prostate Cancer
Brief Title: To Evaluate the Efficacy of TQB3823 Combined With Abiraterone and Prednisone in Metastatic Castration-resistant Prostate Cancer Patientsprednisone Acetate Tablets in Patients With Metastatic Castration-resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor voluntarily terminated the study
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3823-Ib/II-01
Record Dates: First submitted 2022-05-24; First posted 2022-06-06 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
MeSH Terms: interventions — Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3823 tablets + abiraterone acetate tablets + prednisone acetate tablets (Experimental): TQB3823 tablets + abiraterone acetate tablets + prednisone acetate tablets，28 days as a treatment cycle.
  Interventions: Drug: TQB3823 tablets; Drug: Abiraterone acetate tablets; Drug: prednisone acetate tablets

INTERVENTIONS:
Drug: TQB3823 tablets — TQB3823 tablet is an inhibitor of poly ADP-ribose polymerase (PARP).
Drug: Abiraterone acetate tablets — Abiraterone acetate tablet is an inhibitor of cytochrome P450 17（CYP17）
Drug: prednisone acetate tablets — Prednisone acetate tablet is a kind of glucocorticoids

SUMMARY:
This is a phase Ib/II clinical study to explore the safety and efficacy of TQB3823 tablets combined with abiraterone acetate tablets and prednisone acetate tablets in patients with metastatic castration-resistant prostate cancer.

DETAILED DESCRIPTION:
This is a two-phase, open-label Phase Ib clinical trial. The first phase plans to enroll 6-12 patients as two cohorts to explore the safety and of TQB3823 tablets combined with abiraterone and prednisone and the recommended dose of phase II of TQB3823. Subjects involved in cohort one accepts TQB3823 treatment during cycle one and then TQB3823 combined with abiraterone and prednisone from cycle two till the disease progression. The second phase plans to enroll a total of 40-60 subjects, aiming to evaluate the safety and efficacy of TQB3823 tablets combined with abiraterone and prednisone.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18 to 85.
* Subjects with pathologically proven with prostate adenocarcinoma.
* Metastatic disease confirmed by imaging (eg, bone scan and CT/MRI).
* The patient's serum testosterone level at the screening visit was ≤ 1.73 nmol/L (50 ng/dL). Patients who did not undergo bilateral orchiectomy required continued ADT [gonadotropin-releasing hormone analog (LHRHa, agonist/antagonist)] treatment throughout the study period.
* Disease progression during consecutive androgen deprivation therapy (ADT), defined at study entry, as meeting one or more of the following criteria:

  1. At least two consecutive PSA elevations separated by at least 1 week, the last result must be at least 1.0 ng/mL.
  2. Soft tissue lesion progression as assessed by RECIST 1.1 with or without PSA progression.
  3. Bone disease progression assessed by PCWG3, i.e., ≥2 new lesions detected on bone scan, ≥2 new bone lesions other than those previously assessed on reassessment at least 8 weeks later, with ≥2 previously assessed bone lesions still exist, regardless of PSA progression.
* Patients must discontinue all prior cancer therapy (except ADT and bone loss prophylaxis) and have recovered to ≤ Grade 1 or baseline (according to the Common Terminology Criteria for Adverse Events) prior to first dose of all acute toxic effects of prior therapy or surgery Version 5.0 [CTCAE v 5.0]), with the exception of alopecia and peripheral neuropathy, and the washout period since the last prior systemic or radiation therapy was as follows:

  1. At least 4 weeks must have elapsed since enrollment with 5-alpha reductase inhibitors (eg, dutasteride, finasteride), estrogen, and cyproterone.
  2. At least 4 weeks must have elapsed from major surgery or radiation therapy to enrollment。
* Laboratory indicators meet the requirements.

Exclusion Criteria:

* For subjects with brain metastases with symptoms or symptom control for less than 1 month, screening for CNS metastases at baseline is not required unless there are signs and/or symptoms of CNS involvement.
* Subjects who have developed or is currently suffering from other malignancies within 3 years, except for cured skin basal cell carcinoma and cervical carcinoma in situ.
* Subjects who have accepted botanicals (such as saw palmetto) that may lower PSA levels within 4 weeks before the first dose.
* Subjects who have accepted oral targeted drugs within 5 drug half-lives from the first dose (calculated from the end of the last treatment).
* Subjects who have not recovered to ≤ Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 due to the adverse event of prior therapy.
* Subjects who have previously accepted CYP17 enzyme inhibitors (including drugs such as abiraterone, TAK-700, TOK-001, and ketoconazole, ect.,) or second generation androgen receptor inhibitors (including enzalutamide, apalutamide, darolutamide , etc.) (mHSPC, nmCRPC stage).

  1. The study accept patients who received McRpc-based chemotherapy with CYP17 inhibitors other than abiraterone or second-generation androgen receptor inhibitors or paclitaxel for less than 3 months without disease progression, However, 4 weeks or 5 half-life washing out period is required (whichever is longer).
  2. Patients who received abiraterone in the mCRPC phase for less than 3 months and did not progress (no need to stop elution) are allowed in the study, but cannot be enrolled in the phase I cohort of a single drug population in this study.
  3. Patients who received ADT+ paclitaxel chemotherapy, ADT+ 1st generation androgen receptor inhibitors (e.g. Flutamide, bicalutamide, nilutamide, etc.), ADT+ERBT (external radiation therapy) in mHSPC phase will be acceptable in the study, provided that they met the exclusion criteria 2.
* Subjects who receive medications known to be potent inhibitors of cytochrome P450 3A4 (CYP3A4) or potent or moderate inducers and unable to discontinue these medications or switch to another for at least 5 half-lives prior to initiation of study medication different medicines.
* Subjects who suffer from contraindications to prednisone (corticosteroid) use, such as active systemic infection (e.g. bacterial infection requiring intravenous antibiotics at initiation of study treatment, fungal infection, or detectable viral infection requiring systemic therapy ) or viral load (e.g. known HIV positive or known active hepatitis B or C (e.g. hepatitis B surface antigen positive). Screening for contraindications other than HIV/HBV and HCV is not required to determine eligibility.
* Subjects with history of idiopathic pulmonary fibrosis, organizing pneumonia (eg, bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on a chest CT scan during screening.
* Subjects with any chronic condition requiring corticosteroid treatment at doses greater than "Prednisone 5mg, BID";

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Up to 4 weeks
  The relevant adverse reactions occurred within the first cycle
Recommended phase II dose (RP2D) | Up to 8 weeks
  The dose of TQB3823 tablet which is recommended to use during phase II clinical trial
The ratio of subject radiographic progression-free survival for 12 months | For 12 months
  Proportion of subjects without disease progression assessed by radiology within 12 months
Adiographic progression-free survival (rPFS) | Up to 24 months
  rPFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause evaluated by radiological examination

SECONDARY OUTCOMES:
The ratio of subject radiographic progression-free survival for 12 months | For 6 months
  Proportion of subjects without disease progression assessed by radiology within 6 months
The ratio of prostate specific antigen (PSA) reduction | Up to 24 months
  Proportion of subjects with reduction of PSA
Overall response rate (ORR) based on 2014 Lugano | Up to 24 months
  Percentage of participants achieving complete response (CR) and partial response (PR).
Overall survival (OS) | Up to death
  OS defined as the time from randomization until the death from any cause
Clinical benefit rate (CBR) | Up to 24 months
  Proportion of subjects with clinical benefit
Duration of Response (DOR) | Up to 24 months
  The time when the participants first achieved CR or PR to disease progression or death from any cause.
time to bone-related event | Up to 24 months
  Time to progression of bone disease in subjects
Time to PSA progression | Up to 24 months
  Time to raise of PSA in subjects
Peak time (Tmax) | Cycle 1 day 1 and cycle 1 day 28 Before administration, and 1, 2, 4, 6, 8, 11, 12, 24 hours after administration. Cycle 1 day 14 before administration,(each cycle is 28 days)
  The time to peak concentration
Peak concentration (Cmax) | Cycle 1 day 1 and cycle 1 day 28 Before administration, and 1, 2, 4, 6, 8, 11, 12, 24 hours after administration. Cycle 1 day 14 before administration,(each cycle is 28 days)
  Maximum plasma drug concentration
Half-life /T1/2 | Cycle 1 day 1 and cycle 1 day 28 Before administration, and 1, 2, 4, 6, 8, 11, 12, 24 hours after administration. Cycle 1 day 14 before administration,(each cycle is 28 days)
  The time it takes for the drug's concentration in the body to drop by half
Adverse event rate | Baseline up to 96 weeks
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).
Adverse event rate | Baseline up to 24 months
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).

CONTACTS AND LOCATIONS:
Locations (23):
- China (23):
  - The First Hospital of Peking University, Beijing, Beijing Municipality
  - The Southwest Hospitai of Amu, Chongqing, Chongqing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - The Second Hospital of Harbin Medical University, Lanzhou, Gansu
  - Sun Yat-Sun University Cancer Prevertion and Treatment Center, Guangzhou, Guangdong
  - Qingyuan People's Hospital, Qingyuan, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Huadong Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of The Chinese People's Liberation Army Air Force Military Medical University, Xi’an, Shanxi
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Zigong Fourth People's Hospital, Zigong, Sichuan
  - Cancer Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital of Wenzhou Medical Univerity, Wenzhou, Zhejiang